CLINICAL TRIAL: NCT03057496
Title: Wearable Collision Warning Device for Blind and Visually Impaired: Clinical Trial (As Part of: 'Development of a Vision Assistive Device for Veterans With Traumatic Brain Injury-Associated Visual Dysfunctions')
Brief Title: Collision Warning Device for Blind and Visually Impaired
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Alexandra Bowers, Associate Professor of Ophthalmology, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1007377
Record Dates: First submitted 2017-02-14; First posted 2017-02-20 (Actual); Results first posted 2020-12-21 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-01

CONDITIONS: Hemianopia; Hemianopsia; Peripheral Visual Field Defect; Blindness; Retinitis Pigmentosa; Glaucoma
MeSH Terms: conditions — Hemianopsia; Blindness; Retinitis Pigmentosa; Glaucoma

STUDY DESIGN:
Intervention Model Description: The device will operate in two modes: active mode (intervention condition), when it gives warnings and, silent mode (control condition), when it does not give warnings. The device will be programmed to generate a different randomized active/silent schedule for each subject. Participants will not know whether it is in the active or silent mode.
Masking Description: Although this is a single-arm study, participants will be masked in the sense that they will not know whether the device is operating in the active mode (intervention condition), when it gives warnings, or the silent mode (control condition), when it does not give warnings. The device will be programmed to generate a different randomized active/silent schedule for each subject. The investigator conducting the statistical analyses will also be masked as to whether the device was in the active or silent mode
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental): Participants will use the collision warning device as much as possible for about one month during everyday activities, when walking indoors and outdoors.
  Interventions: Device: Collision warning device

INTERVENTIONS:
Device: Collision warning device — The collision warning device is a pocket-sized, electronic system that includes a micro-computer, a clip-on miniature camera, a gyro-sensor, an accelerometer, and a rechargeable battery, all contained within a shoulder bag. It is about the size of a smart phone. When a potential collision is detected by the device it emits a warning to the user, either in the form of an audible beep or a tactile warning through bracelets worn on the wrist. The time to collision will be coded in both the auditory and tactile domains. The device is designed to only give warnings about high risk collisions, so the users will not be continually bombarded by warnings for every potential collision object in the environment.

SUMMARY:
This study evaluates a novel collision warning device to help people with severe vision impairment or blindness avoid collisions with obstacles. The main hypothesis to be tested is that the device reduces the number of collisions with obstacles in everyday activities.

DETAILED DESCRIPTION:
Participants with blindness or severe visual field loss (hemianopia or tunnel vision) will be trained to use a collision warning device that alerts them to impending collisions. Participants will use the device at home during everyday mobility for about 1 month. The device is designed to supplement existing mobility devices, such as a long cane or dog guide. The device will provide warnings about potential collisions with mid- or high-level obstacles (which are typically not detected by a long cane).

ELIGIBILITY:
Inclusion Criteria:

* Blindness (or very limited vision with visual acuity no better than "counting fingers"),
* Or severe peripheral field loss / tunnel vision (≤ 40° remaining visual field) with visual acuity of at least 20/200,
* Or homonymous hemianopia with visual acuity of at least 20/200;
* Able to walk independently either with or without mobility aids such as a long cane or guide dog (but without the aid of a sighted guide);
* Reports at least minor bumps or collisions within the last 3 months;

Exclusion Criteria:

* Currently participating in a mobility training program
* Diagnosed dementia
* Significant cognitive decline
* Participants with hemianopia will be excluded if they have hemianopia for less than 3 months and/or have spatial neglect

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Bowers, PhD, Principal Investigator — Schepens Eye Research Institute, Mass Eye and Ear; Gang Luo, PhD, Principal Investigator — Schepens Eye Research Institute, Mass Eye and Ear
Locations (1):
- Schepens Eye Research Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pundlik S, Baliutaviciute V, Moharrer M, Bowers AR, Luo G. Data Acquisition, Processing, and Reduction for Home-Use Trial of a Wearable Video Camera-Based Mobility Aid. Transl Vis Sci Technol. 2020 Jun 11;9(7):14. doi: 10.1167/tvst.9.7.14. eCollection 2020 Jun. PMID 32832221
- [Derived] Pundlik S, Baliutaviciute V, Moharrer M, Bowers AR, Luo G. Home-Use Evaluation of a Wearable Collision Warning Device for Individuals With Severe Vision Impairments: A Randomized Clinical Trial. JAMA Ophthalmol. 2021 Sep 1;139(9):998-1005. doi: 10.1001/jamaophthalmol.2021.2624. PMID 34292298

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between January 2018 and May 2019 via referrals from the Carroll Center for the Blind, the Massachusetts Commission for the Blind and practitioners at vision rehabilitation clinics in the Greater Boston area, and via a pool of volunteers who had previously participated in studies in our lab.
Groups:
- Silent and Active Mode: During the period of home-use of the device, all participants experienced both the silent and active modes on a random schedule. Thus participant flow was the same for silent and active modes and is described for all participants together.
Period: Overall Study
Arm/Group | Silent and Active Mode
Started | 49
Started Home-use Trial | 36
Completed | 31
Not Completed | 18
Not completed — Withdrawal by Subject | 8
Not completed — Lost to Follow-up | 5
Not completed — Did not use device during home trial | 3
Not completed — Device failure | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes only those subjects who completed the one-month period of device use and had data successfully recorded by the device.
Groups:
- Silent and Active Mode: During the period of home-use of the device, all participants experienced both the silent and active modes on a random schedule. Thus the baseline measures are the same for active and silent modes (as it was the same participants for both modes) and are reported together.
Arm/Group | Silent and Active Mode
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: Years] | 61 [25 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 18
  More than one race | 1
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 31
Habitual mobility aid [Count of Participants; unit: Participants]
  Long cane | 28
  Guide dog | 3
Cause of vision impairment [Count of Participants; unit: Participants]
  Retinitis Pigmentosa | 8
  Retinopathy of prematurity | 5
  Other | 15
  Unknown | 3
Vision impairment onset [Count of Participants; unit: Participants]
  At birth | 17
  Adult | 14
Duration of vision loss [Median (Full Range); unit: years] | 38 [5 to 73]
Amount of vision [Count of Participants; unit: Participants]
  No light perception | 11
  Light perception | 8
  Better than light perception | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Collision Incidents (All Contacts)
Description: Collision incidents recorded by the device in everyday use, including long cane contacts and body contacts with surrounding objects in the environment.
Time Frame: During the one-month period of device use
Population: The device switched between active and silent modes on a random schedule so data about collision incidents were available for each subject for both conditions
Measure: Median (Inter-Quartile Range); unit: Rate (contacts per 100 hazards per hour)
Groups:
- Silent Mode: Participants used the collision warning device as much as possible for about one month during everyday activities, when walking indoors and outdoors. The device switched between silent and active mode on a random schedule. In the silent mode the device detected potential collisions but did not provide any active warnings to the users.
- Active Mode: Participants used the collision warning device as much as possible for about one month during everyday activities, when walking indoors and outdoors. The device switched between silent and active mode on a random schedule. In the active mode the device detected potential collisions and gave active warnings to the users via vibro-tactile wristbands.
Arm/Group | Silent Mode | Active Mode
Number analyzed (Participants) | 31 | 31
Rate (contacts per 100 hazards per hour) | 13.79 [7.28 to 24.29] | 9.26 [6.56 to 14.96]
Statistical Analysis 1: Comparison: Silent Mode vs Active Mode; A within-subject comparison was performed. Each subject included in the analysis used the device in both the active and the silent mode. Comparison was between the two device operating modes. The null hypothesis was that there was no difference in the rate of contacts between active and silent modes; Test type: Superiority; p < 0.001, Mixed Models Analysis — Since the outcome (contacts) represented over-dispersed count data and there were repeated measurements per subject, a generalized mixed effects model with a negative binomial family was used with each subject treated as a random intercept; Fixed factors were included in the model to account for factors other than device operating mode that might affect collision rates; Rate ratio = 0.627, 95% CI 2-sided [0.536 to 0.734], Standard Error of Mean 0.08 — Silent mode is the denominator for the rate ratio

2. Secondary Outcome: Number of Body Contacts
Description: Collision incidents with body contacts recorded by the device
Time Frame: During the one-month period of device use
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Rate (contacts per 100 hazards per hour)
Arm/Group | Silent Mode | Active Mode
Number analyzed (Participants) | 31 | 31
Rate (contacts per 100 hazards per hour) | 1.13 [0.45 to 3.08] | 1.09 [0.3 to 1.97]

3. Secondary Outcome: Device Questionnaire
Description: Questionnaire addressing participants' experiences of using the device. Scores were on a 5-point rating scale (1 to 5) with higher scores representing a better score. Questions were grouped into four main categories: i) overall satisfaction, ii) comfort, iii) mobility benefit, and iv) ease of operation. An average score was computed for questions within each category.
Time Frame: During the one-month period of device use
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Silent and Active Mode: Since participants did not know when the device was in either the silent or the active mode, it was not possible for them to answer questions specific to each mode. The questionnaire was completed after using the device for one month and therefore represents ratings of the device for the whole duration of the trial including both active and silent operating modes.
Arm/Group | Silent and Active Mode
Number analyzed (Participants) | 30
scores on a scale
  Overall satisfaction | 3.68 (0.74)
  Comfort | 4.08 (0.53)
  Mobility benefit | 3.05 (1.08)
  Ease of operation | 3.96 (0.49)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the one-month period when subjects were using the device.
Description: A brief questionnaire was administered to each subject by telephone each week during the one-month period of device use to check on how much they were using the device and whether they had encountered any difficulties. One question specifically asked whether the subject had experienced any adverse events.
Groups:
- Silent and Active Mode: During the period of home-use of the device, all participants experienced both the silent and active modes on a random schedule. Neither the subject nor the researcher recording adverse events knew whether the device was in silent or active mode at the time when an event occurred, thus the adverse events are reported for all participants and both modes together.
Arm/Group | Silent and Active Mode
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 6/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silent and Active Mode (N=36)
Minor contact with object in the environment (General disorders) | 6 (8) — A minor contact, brushing against or bumping into an object (e.g., bushes, overhanging branches) in the environment when walking

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-01-26): https://cdn.clinicaltrials.gov/large-docs/96/NCT03057496/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT03057496/Prot_SAP_002.pdf